CLINICAL TRIAL: NCT05804292
Title: Psychometric Proprieties and Validation of Self-report Measures of Eating Behaviors in Persons With Obesity and the General Population in Italy.
Brief Title: Psychometric Proprieties and Validation of Self-report Measures of Eating Behaviors
Acronym: Valid-OB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 03C020
Record Dates: First submitted 2023-03-15; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Eating Disorders
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Community sample: Questionnaires administration
  Interventions: Other: Questionnaire administration
- Subjects with obesity and comorbid eating disorder: Questionnaires administration
  Interventions: Other: Questionnaire administration
- Subjects with obesity without comorbid eating disorder: Questionnaires administration
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — Questionnaire administration

SUMMARY:
Obesity is a global epidemic and a major contributor to some of the leading causes of death.

Although research on overweight and obesity is constantly increasing, to date, in the Italian panorama, there is a lack of (A) rigorous psychological measurement tools of obesity-related constructs and (B) analysis of the relationships between constructs (and indicators) involved in the development and maintenance of overweight and obesity.

The present study aims to examine the psychometric properties of the main questionnaires for the assessment of eating behaviors in 3 groups of subjects (1) the general population (control group); (2) subjects with obesity without a comorbid diagnosis of an eating disorder; (3) subjects with obesity and a comorbid diagnosis of an eating disorder.

DETAILED DESCRIPTION:
Participants were selected in the main rehabilitation centers for the treatment of obesity and eating disorders (sample of subjects with obesity) and through an online survey (community sample). The survey lasted about 30 minutes and - together with selected demographic and biomedical information - required the completion of the following self-report measures: the Binge Eating Scale (BES); the Modified Yale Food Addiction Scale version 2 (mYFAS 2.0); the Repetitive eating questionnaire (Rep-EAT); the Measure of Eating Compulsivity (MEC); the Addiction-like Eating Behavioural Scale (AEBS); the Three Factor Eating Questionnaire 18 (TFEQ-18); the Eating Disorders Examination Questionnaire-Short Form (EDEQ-SF); the Palatable Eating Motive Scale (PEMS); the Weight Sigma Questionnaire (WSSQ); the Emotional Eating Scale (EES); the Somatic Symptom Scale 8 (SSS8).

Before administration, all questionnaires were first translated from English (their original language) to Italian by two bilingual translators, independently - then back-translated into English by another independent translator whose mother tongue was English to ensure equivalence between the translations. Following, a purposive sample of respondents was asked to fill in the final version of each measure in order to assess its items' comprehensibility.

In order to avoid halo effects, the questionnaires were presented to the subject in random order.

The responders could withdraw the administration at any time, and contact a psychologist independent from the study in case of perceived emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2 (clinical sample)
* Diagnosis of an eating disorder (clinical sample)
* age range 18-75 years
* Italian mother tongue
* written and informed consent to participate

Exclusion Criteria:

* visual impairing
* neurological problems
* alcohol/drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with obesity with/without an eating disorder AND the general population (non clinical)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Binge Eating | Baseline
  Score on the Binge Eating Scale. Each question has 3-4 separate responses assigned a numerical value. The score range is from 0-46: Non-binging; less than 17; Moderate binging; 18-26; Severe binging; 27 and greater
Food Addiction | Baseline
  Scored on the Modified Yale Food Addiction Scale version 2 and at the Addiction-like Eating Behavioural Scale The "symptom count" score, ranging from 0 to 7, that reflects the number of addiction-like criteria endorsed was applied

CONTACTS AND LOCATIONS:
Overall Officials: Giada Pietrabissa, PhD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No